CLINICAL TRIAL: NCT04996589
Title: Exploring the Potential of Finger Prick Blood for Assessment of BIOmarkers for LOw Grade Inflammation and CVD Risk
Acronym: BIOLOGIC
Status: Completed | Type: Observational
Sponsor: Wageningen University and Research (Other)
Responsible Party: Principal Investigator, Diederik Esser, Clinical Trial Coordinator, Wageningen University and Research
Other Study IDs: NL76207.091.20
Record Dates: First submitted 2021-07-27; First posted 2021-08-09 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Biomarker
Keywords: LPS; biomarker; finger prick test; postprandial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Venous blood samples and blood collected via finger pricks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lean subjects: BMI 18.5-22
- Obese subjects: BMI>30

SUMMARY:
There are currently no minimally invasive techniques for the measurement of lipopolysaccharide (LPS) and Apo-B48 that can be used in samples collected in field settings. In this project we want to explore whether postprandial assessment of biomarkers LPS and ApoB48 in blood withdrawn with a finger prick test can be used as marker for low grade inflammation and risk factor for CVD.

The primary objectives of this pilot study are to a) determine whether postprandial LPS and ApoB48 levels can be assessed in finger prick blood of both lean subjects and obese subjects; and b) compare postprandial LPS and ApoB48 levels assessed in venous blood and blood collected through a finger prick test.

This study is an observational pilot study in which postprandial LPS and ApoB48 will be assessed before and after ingestion of a high fat load in 5 lean and 5 obese subjects in the age range 18-70 years.

Samples will be collected under fasting conditions and in response to a high fat challenge test (1, 2, 4 and 6 hours post ingestion).

The risks for participation are very small if not negligible. No adverse effects of the high fat challenge were reported previously. Consumption of high amounts of saturated fat may cause some GI discomfort. Blood sampling will be performed via a cannula and the insertion can be a painful and may cause a bruise. Finger prick might also give a short pain sensation and small bruises. The amount of blood that is drawn from participants is relatively small (total 37.5 ml) and is therefore within acceptable limits. There are no direct benefits for the participants. In the BIOLOGIC study we include both lean subjects and obese subjects as we expect differences in postprandial responses related to differences in chylomicron production and LPS levels. Therefore it is important to explore these biomarkers in both target groups. This study can therefore be regarded as group-related, non-therapeutic research.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Living in the surroundings of Wageningen (max. 25 km)
* Stable body weight for past 6 months
* Suitable veins for insertion of cannula
* BMI 18.5-22 kg/m2 (lean subjects)
* BMI ≥ 30 kg/m2 (obese subjects)

Exclusion Criteria:

* Use of cholesterol-lowering medication (e.g. statins)
* Use of diabetes medication (e.g. insulin, metformin)
* Use of antibiotics or anti-inflammatory medication (e.g. NSAIDS such as ibuprofen)
* Known allergy for any of the food components used in the study (milk, cream, sugars)
* Blood clotting disorders
* Current smokers
* Alcohol consumption of > 21 units per week
* Participation in another clinical trial at the same time
* Being an employee of Wageningen Food & Biobased Research

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In the current study we aim to include 5 lean subjects and 5 obese subjects. We expect different biomarker responses to a high fat load between these groups of subjects and therefore it is relevant to explore whether the proposed biomarkers are valid in both sub population groups.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
LPS_B1 | Baseline
  Serum levels LPS venous blood samples under fasting conditions
ApoB48_B1 | Baseline
  Serum levels ApoB48 venous blood samples under fasting conditions
LPS_B2 | Baseline
  Serum levels LPS finger prick blood under fasting conditions
ApoB48_B2 | Baseline
  Serum levels ApoB48finger prick blood under fasting conditions
LPS1-1 | 1 hour post ingestion
  Serum levels LPS venous blood samples after high-fat shake intake
ApoB48_1-1 | 1 hour post ingestion
  Serum levels ApoB48 venous blood samples after high-fat shake intake
LPS1-2 | 1 hour post ingestion
  Serum levels LPS finger prick blood after high-fat shake intake
ApoB48_1-2 | 1 hour post ingestion
  Serum levels ApoB48 finger prick blood after high-fat shake intake
LPS2-1 | 2 hours post ingestion
  Serum levels LPS venous blood samples after high-fat shake intake
ApoB48_2-1 | 2 hours post ingestion
  Serum levels ApoB48 venous blood samples after high-fat shake intake
LPS2-2 | 2 hours post ingestion
  Serum levels LPS finger prick blood after high-fat shake intake
ApoB48_2-2 | 2 hours post ingestion
  Serum levels ApoB48 finger prick blood after high-fat shake intake
LPS4-1 | 4 hours post ingestion
  Serum levels LPS venous blood samples after high-fat shake intake
ApoB48_4-1 | 4 hours post ingestion
  Serum levels ApoB48 venous blood samples after high-fat shake intake
LPS4-2 | 4 hours post ingestion
  Serum levels LPS finger prick blood after high-fat shake intake
ApoB48_4-2 | 4 hours post ingestion
  Serum levels ApoB48 finger prick blood after high-fat shake intake
LPS6-1 | 6 hours post ingestion
  Serum levels LPS venous blood samples after high-fat shake intake
ApoB48_6-1 | 6 hours post ingestion
  Serum levels ApoB48 venous blood samples after high-fat shake intake
LPS6-2 | 6 hours post ingestion
  Serum levels LPS finger prick blood after high-fat shake intake
ApoB48_6-2 | 6 hours post ingestion
  Serum levels ApoB48 finger prick blood after high-fat shake intake

SECONDARY OUTCOMES:
LBP_B | Baseline
  Plasma LBP levels in venous blood samples collected under fasting conditions
LBP_1 | 1 hour post ingestion
  Plasma LBP levels in venous blood samples after high-fat shake intake
LBP_2 | 2 hours post ingestion
  Plasma LBP levels in venous blood samples after high-fat shake intake
LBP_4 | 4 hours post ingestion
  Plasma LBP levels in venous blood samples after high-fat shake intake
LBP_6 | 6 hours post ingestion
  Plasma LBP levels in venous blood samples after high-fat shake intake
sCD14_B | Baseline
  Plasma sCD14 levels in venous blood samples collected under fasting conditions
sCD14_1 | 1 hour post ingestion
  Plasma sCD14 levels in venous blood samples after high-fat shake intake
sCD14_2 | 2 hours post ingestion
  Plasma sCD14 levels in venous blood samples after high-fat shake intake
sCD14_4 | 4 hours post ingestion
  Plasma sCD14 levels in venous blood samples after high-fat shake intake
sCD14_6 | 6 hours post ingestion
  Plasma sCD14 levels in venous blood samples after high-fat shake intake

CONTACTS AND LOCATIONS:
Locations (1):
- Stichting Wageningen Research, Wageningen, Gelderland, Netherlands